CLINICAL TRIAL: NCT02850809
Title: Evaluation of the Efficacy of Radiofrequency Ablation in the Treatment of Renal Tumors: Prospective Observational Study
Brief Title: Evaluation of the Efficacy of Radiofrequency in the Treatment of Renal Tumors
Acronym: RF-REIN
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Ministry for Health and Solidarity, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2010/08
Record Dates: First submitted 2016-07-25; First posted 2016-08-01 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Renal Cell Carcinoma
Keywords: radiofrequency ablation; complications
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients: Treated by percutaneous image-guided radiofrequency for renal tumor

SUMMARY:
Multi-institutional registry on a cohort of 310 patients with biopsy-proven renal cell carcinoma treated by Radiofrequency ablation. All patients will be included consecutively and retrospectively in all centers to obtain the required number of patient followed during 5 years.

DETAILED DESCRIPTION:
Radiofrequency ablation (RFA) of renal cell carcinoma (RCC) is actually used in elderly patients with small renal tumors (diameter ≤ 4 cm) and presenting a high risk of surgery (due to co-morbidity) and/or reduced renal function. RFA is a minimally invasive technique, considered as an alternative to surgery to limit morbidity and to preserve kidney function. The technique is well known and has proven his efficacy for the treatment of small tumors.

An enlargement of the indications of RFA to patient without contra-indication to surgery will depend on the efficacy of the technique.

The main objective of the study is to evaluate the local efficacy of the ablation based on the technical success, and on the evaluation of local cancer recurrence over 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with percutaneous RFA
* Patient with diagnosis of renal masses with a maximum of 3 masses treated during the ablation
* The diameter of the tumor must be ≤ 40 mm, characterized by CT-scan or MRI
* The histology of the tumor must be biopsy-proven or the patient must have previous surgical ablation of renal tumor (ipsi or contralateral)

Exclusion Criteria:

* Patient treated by surgery or laparoscopy
* Benign tumors
* No histological diagnosis (no biopsy or no previous treated renal carcinoma)
* Patient having secondary malignant sites, ganglions or visceral metastatic cells or endo-venous extend at the time of RFA
* Patient having a diagnosis of primary or secondary extra-renal tumor location and not into remission
* Patients treated with antiangiogenic drugs during the 6 months prior RFA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population concerned by the study consists in patients treated by percutaneous image-guided radiofrequency for renal tumor. The treated tumors have a diameter ≤ 4 cm characterized by computed tomography (CT) or Magnetic resonance imaging (MRI).
Sampling Method: Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2010-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Rate of local efficacy of RFA treatment | 60 months after the RFA treatment (D0)

SECONDARY OUTCOMES:
Overall success | At 60 months after the RFA treatment (D0)
No recurrence of RCC | At 60 months after the RFA treatment (D0)
Tolerance of the treatment | At D0, 48 hours, 6, 12, 24, 36, 48 and 60 months after the RFA treatment (D0)

CONTACTS AND LOCATIONS:
Overall Officials: Paul PEREZ, MD, Study Chair — University Hospital Bordeaux, France; Nicolas GRENIER, Prof, Principal Investigator — University Hospital Bordeaux, France
Locations (8):
- France (8):
  - CHU de Bordeaux - Pellegrin, Bordeaux
  - CHU de Grenoble, Grenoble
  - CHRU de Lille - Hôpital Claude HURIEZ, Lille
  - Hospices Civils de Lyon, Lyon
  - Assistance Publique - Hôpitaux de Marseille, Marseille
  - Assistance Publique - Hôpitaux de Paris (AP-HP) - Hopital Necker, Paris
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Hopital de Rangueil, Toulouse